CLINICAL TRIAL: NCT02926924
Title: Prophylactic Application of an Incisional Wound Vac to Prevent Wound
Brief Title: Prophylactic Application of an Incisional Wound Vac to Prevent Wound Complications in Obese Spine Surgery Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Rakesh Patel, Clinical Assistant Professor, Orthopaedic Surgery, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HUM00050885
Record Dates: First submitted 2016-10-04; First posted 2016-10-06 (Estimated); Results first posted 2025-04-11 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-03

CONDITIONS: Spine Surgery; Wounds Vac
MeSH Terms: interventions — Negative-Pressure Wound Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Wound Vac (Active Comparator): Wound vac
  Interventions: Device: Wound Vac
- Standard Dressing (Active Comparator): Standard Dressing
  Interventions: Other: Standard Dressing

INTERVENTIONS:
Device: Wound Vac — a therapeutic technique using a vacuum dressing to promote healing in acute or chronic wounds and enhance healing of first and second degree burns.
  Other Names: Negative pressure therapy
  Arms: Wound Vac
Other: Standard Dressing — standard dressing with drain tube and bandage
  Arms: Standard Dressing

SUMMARY:
This is a prospective randomized study evaluating the use of a prophylactic incision wound vac dressing, applied in the OR, on patients undergoing posterior spine surgery with a BMI>35. Patients are randomized in the operating room to normal postoperative dressing vs. vac dressing. The vac dressing would be left on for 72 hours postoperatively. In the interim, the patients' postoperative care can proceed as usual. Our primary outcomes will be antibiotics or return trip needed to the operating room for wound related complications.

The patients only intervention would be the application of an incisional wound vac. The will be no change in the patients postoperative protocol otherwise. This procedure is noninvasive.

ELIGIBILITY:
Inclusion Criteria:

* Be scheduled to have posterior spine surgery (inpatient procedures only).
* Have a BMI greater than or equal to 35.

Exclusion Criteria:

* BMI less than 35
* Previous spine infection
* Intraoperative dural tear

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2011-08-01 (Actual); Primary Completion 2015-01-15 (Actual); Study Completion 2015-01-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rakesh Patel, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of 68 participants consented, 2 were excluded by PI decision for coming from another site and their data is not accessible for inclusion in any analyses. Of the remaining 66, data for 26 was irretrievably lost and cannot be provided. One participant in the standard group subsequently participated in the wound vac group (without an additional consent required), as is shown by the milestone listed below.
Period: Overall Study
Arm/Group | Standard Dressing | Wound Vac
Started (Started here means randomized to this arm and began in this arm and for whom data is recoverable/verifiable.) | 19 | 21
S.D. First Then After a Subsequent Surgery Participated in WV Without Reconsent or Re-randomization | 1 | 0 (The participant shown in this milestone in the standard dressing arm did in fact participate in the wound vac arm after a second surgery, but is shown here as "0" because that person was not initially randomized to this arm, and therefore doesn't show in the 21 "started")
Completed | 19 | 20
Not Completed | 0 | 1
Not completed — withdrawal - reason unknown | 0 | 1

BASELINE CHARACTERISTICS:
Population: 28 participants' data (2 from elsewhere and 26 from Michigan) was lost and their baseline data is not included. The individual who began in the standard dressing group and then subsequently participated in the wound vac group is only represented in the standard dressing group for baseline characteristics analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Dressing | Wound Vac | Total
Number analyzed (Participants) | 19 | 21 | 40
Age, Continuous [Mean (Full Range); unit: years] | 55 [35 to 73] | 56 [38 to 79] | 55.2 [35 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 12 | 25
  Male | 6 | 9 | 15
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 19 | 21 | 40

OUTCOME MEASURES:

1. Primary Outcome: Count of Patients With Post Operative Infection
Description: Count of Patients with Post operative infection requiring return to operating room or prolonged treatment of antibiotics
Time Frame: 6 weeks post surgery
Population: 22 are shown in the wound vac arm because of the one participant whose first surgery was with standard dressing and subsequently participated in the wound vac arm after a second surgery.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Dressing | Wound Vac
Number analyzed (Participants) | 19 | 22
Participants
  readmission | 4 | 2
  prolonged antibiotic use | 5 | 3

ADVERSE EVENTS:
Time Frame: 6 weeks after surgery
Description: The only adverse events that were collected were extended antibiotic use and rehospitalization. So the 0s listed in "other adverse events" is simply a statement of what data was collected, but not an assurance that no non-serious adverse events occurred.
  Systematic assessment was performed simply by a records review pulling for those two items: extended antibiotic use and rehospitalization.
Arm/Group | Standard Dressing | Wound Vac
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/22
Serious Adverse Events (participants affected / at risk) | 4/19 | 2/22
Other Adverse Events (participants affected / at risk) | 5/19 | 3/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard Dressing (N=19) | Wound Vac (N=22)
Readmission to Hospital (Surgical and medical procedures) | 4 | 2 — required return trip to the operating room for what was found to be a suture abscess
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard Dressing (N=19) | Wound Vac (N=22)
prolonged antibiotic use required (Infections and infestations) | 5 | 3

LIMITATIONS AND CAVEATS:
This small study was intended to be a pilot. Without a larger population, results should not be seen as generalizable.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes